CLINICAL TRIAL: NCT02913755
Title: Improving Treatment Motivation and Self-awareness in People With Moderate to Severe Acquired Brain Injury (ABI)
Brief Title: Motivation and Self-awareness in Acquired Brain Injury (ABI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Brain Injury Rehabilitation Trust (Other)
Responsible Party: Principal Investigator, Hamish J McLeod PhD CPsychol, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16/WS/0232
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Repeated viewing of a short Preparatory video about ABI rehabilitation; viewed every 2-3 days over a 4 week period
  Interventions: Behavioral: Preparatory video
- Lagged Control Group (Active Comparator): 2 week period of treatment as usual followed by repeated viewing of a short Preparatory video about ABI rehabilitation; viewed every 2-3 days over a 4 week period
  Interventions: Behavioral: Preparatory video

INTERVENTIONS:
Behavioral: Preparatory video — 5 minute Preparatory video to increase motivation, awareness and engagement in ABI rehabilitation

SUMMARY:
Acquired Brain Injury (ABI) is damage to the brain caused by a head injury or illness/disease such as stroke or aneurysm. ABI is often associated with poor awareness into ongoing symptoms of damage to the brain, which can be cognitive, physical, and psychological. A multi-disciplinary rehabilitation programme is recommended to help with such symptoms. However, without self-awareness of difficulties, people with ABI can have poor motivation to take part. The study aims to discover whether showing people a short 'preparatory' video about ABI rehabilitation has an effect on self-awareness, and their motivation to take part in rehabilitation offered to them.

The study also aims to investigate the feasibility of using the preparatory video on a larger scale across inpatient ABI rehabilitation, by exploring whether staff find delivering the video easy to incorporate into routine practice.

People invited to take part in the study will be recruited from a specialist inpatient brain injury rehabilitation unit (BIRT).

People who are approached will be given information about what the study will involve, and can choose not to take part.

Each participant will be asked to fill out a series of questionnaires. They will then be supported by staff to watch a short video every two/three days, over four weeks. Half of the participants will be shown the video right away, while the other half will wait two weeks, to allow for comparisons between the groups. The video will aim to improve understanding of the kinds of emotional and/or practical difficulties they may be experiencing, and will inform participants about what rehabilitation might be like. After they have regularly watched the video for four weeks both sets of participants will be asked to complete another set of questionnaires, and the staff will be asked to complete an evaluation of how they found delivering the video.

DETAILED DESCRIPTION:
The study will be a repeated-measures design, with a lagged control group, allowing within- and between-subjects analysis. The primary outcome variable is motivation for rehabilitation (Motivation for traumatic brain injury rehabilitation questionnaire - MOT-Q). Secondary measures include measures of awareness (Awareness Questionnaire - AQ) and behaviour change (The Pittsburgh Rehabilitation Participation Scale - PRPS, and participation statistics). Tertiary outcomes are the assessment of the feasibility of the preparatory material as an intervention, completed by BIRT staff (Structured Assessment of Feasibility measure - SAFE).

Primary participants will be recruited from a brain injury inpatient unit in Glasgow provided by Brain Injury Rehabilitation Trust (BIRT), and information recorded from case notes. This will include demographics, information about the brain injury, a cognitive profile, and participation statistics relating to attendance in their BIRT rehabilitation programme. Primary and secondary outcome measures (MOT-Q, AQ) will be completed.

Participants will then be randomly stratified (by time since admission, and motivation for rehabilitation) into two groups; intervention and control. All participants will view the preparatory video in a 1:1 delivery by a member of BIRT staff every 2-3 days over a period of 4 weeks, with the control group on delayed exposure of 2 weeks. During the delay period, the control group will continue to receive routine care from BIRT rehabilitation staff. BIRT staff will record the number of videos scheduled and watched by each participant.

Primary and secondary outcome measures (MOT-Q, AQ) will be completed by inpatient participants again mid- and post-trial to allow exploration of effects by within-group comparisons, and between-group comparison with control group.

Staff participants will complete the AQ and PRPS pre- and post-trial. Routine participation statistics recorded by staff will be gathered pre- and post-trial. Additionally, staff will evaluate of the feasibility of delivering the protocol, by completing the SAFE questionnaire post-trial.

ELIGIBILITY:
Inclusion Criteria:

* current inpatients with moderate-severe ABI (i.e. damage to the brain's physiology caused by an external force or pathophysical damage resulting from non-degenerative organic factors such as stroke, encephalitis, aneurysm, neurological disease)
* aged >18 years
* capacity to give consent

Exclusion Criteria:

* communication difficulties that might affect ability to consent to or understand/comply with test procedures
* severe mental illness or challenging behaviour that would prevent meaningful participation in the study
* a discharge date within the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Motivation for traumatic brain injury rehabilitation | Change from baseline to 4 weeks
  Score from Motivation for traumatic brain injury rehabilitation questionnaire - MOT-Q

SECONDARY OUTCOMES:
Awareness | Change from baseline to 4 weeks
  Score from Awareness Questionnaire - AQ
Behaviour change | Change from baseline to 4 weeks
  Score from Pittsburgh Rehabilitation Participation Scale - PRPS
Feasibility | 4 weeks
  Score from Structured Assessment of Feasibility measure (SAFE)
Feasibility of intervention delivery | 4 weeks
  Percentage of scheduled videos delivered to each participant
Rehabilitation participation | 4 weeks
  Number of rehabilitation sessions offered/attended/refused

CONTACTS AND LOCATIONS:
Overall Officials: Hamish McLeod, Principal Investigator — University of Glasgow
Locations (1):
- Brain Injury Rehabilitation Trust, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No